CLINICAL TRIAL: NCT06452550
Title: Multimodal MRI-based Neurophenotype Reflecting Brain-gut Interactions to Predict Intestinal Disease Progression in Patients With Crohn's Disease
Brief Title: Neurophenotype Predicts CD Disease Progression
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xuehua Li, associate chief physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: 82070680
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Radiomics; Multi-omics
Keywords: Abdominal MRI; Magnetic Resonance Imaging; Crohn's disease; Brain/gut interaction
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn's disease patients with no-to-mild inflammation: On MR enterography, the Magnetic Resonance Index of Activity (MaRIA) and Magnetic Resonance Enterography Global Score (MEGS) were used to characterize intestinal inflammation by assessing intramural and extramural lesions in both the small and large intestines. In ileocolonoscopy, the Simplified Endoscopic Activity Score for Crohn's Disease (SES-CD) was used to quantify mucosal or luminal lesions from the terminal ileum to the colorectum. Both modalities were used to classify patients with no-to-mild or moderate-to-severe inflammation. We defined patients as having moderate-to-severe inflammation when at least two of the following criteria were met: (1) MaRIA≥11; (2) MEGS≥ 10 for the small bowel or MEGS≥12 for the colon; or (3) SES-CD≥11. Otherwise, patients were categorized as having no-to-mild inflammation.
  Interventions: Diagnostic Test: Logistic regression (LR) prediction models
- Crohn's disease patients with moderate-to-severe inflammation: On MR enterography, the Magnetic Resonance Index of Activity (MaRIA) and Magnetic Resonance Enterography Global Score (MEGS) were used to characterize intestinal inflammation by assessing intramural and extramural lesions in both the small and large intestines. In ileocolonoscopy, the Simplified Endoscopic Activity Score for Crohn's Disease (SES-CD) was used to quantify mucosal or luminal lesions from the terminal ileum to the colorectum. Both modalities were used to classify patients with no-to-mild or moderate-to-severe inflammation. We defined patients as having moderate-to-severe inflammation when at least two of the following criteria were met: (1) MaRIA≥11; (2) MEGS≥ 10 for the small bowel or MEGS≥12 for the colon; or (3) SES-CD≥11. Otherwise, patients were categorized as having no-to-mild inflammation.
  Interventions: Diagnostic Test: Logistic regression (LR) prediction models

INTERVENTIONS:
Diagnostic Test: Logistic regression (LR) prediction models — Logistic regression model was used to establish a model to distinguish different levels of intestinal inflammation.

SUMMARY:
The goal of this observational study is aimed to develop a novel multimodal neuroimaging-based model to characterize the neurophenotype of Crohn's Disease patients and assess its ability for predicting disease progression, using multiomics data to interpret the model.

Participants will be followed-up of at least six months for patients without disease progression to assess the relationship between neurophenotype and intestinal outcomes.

DETAILED DESCRIPTION:
Brain-gut axis plays a crucial role in the pathogenesis of Crohn's disease (CD); however, CD neurophenotype and its impact on intestinal disease progression remain unclear. We aimed to develop a novel multimodal neuroimaging-based model to characterize the neurophenotype of CD patients and assess its ability for predicting disease progression, using multiomics data to interpret the model. This study enrolled CD patients who underwent baseline testing (including neuroimaging, psychological scales, MR enterography, and ileocolonoscopy) and faecal/blood samples collection. The neurophenotypes of patients were characterized using a neuroimaging-based model. The predictive ability of neurophenotype model for disease progression was evaluated using Cox regression analysis. Multiomics data (including faecal microbiome, faecal/blood metabolomics, intestinal permeability, blood-brain-barrier permeability, and blood neurotransmitter levels) were used to elucidate how neurophenotypes reflect brain-gut interactions.

ELIGIBILITY:
Inclusion Criteria:

* (a) CD patients aged 18-45 years; (b) the completion of multimodal brain MRI and administration of psychological questionnaires; (c) MR enterography (MRE), ileocolonoscopy, and blood or faecal samples, collection within one week of brain MRI; (d) a follow-up of at least six months for patients without disease progression; and (e) right-handedness.

Exclusion Criteria:

* (a) recent use of antibiotics, probiotics, or prebiotics within three months prior to inclusion; (b) history of neurosurgery, cerebrovascular disease, or brain trauma; (c) use of central nervous system drugs or antidepressants within three months prior to inclusion; (d) identification of brain lesions on MR scan; (e) claustrophobia; or (f) presence of metal implants.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study included adult patients aged 18 to 45 with Crohn's disease (CD) who were admitted to the First Affiliated Hospital of Sun Yat-sen University between May 2021 and June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The area under the ROC curve (AUC) to assess the performance of diagnostic model | 6 months
  After baseline brain MRI scanning, patients were followed up.

CONTACTS AND LOCATIONS:
Overall Officials: Xuehua Li, Principal Investigator — Sun Yat-sen University First Affiliated Hospital Department of Radiology
Locations (1):
- XploreMET v3.0 system, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Disclosure is subject to application